CLINICAL TRIAL: NCT02216357
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Trial to Determine the Safety of Oral Ifetroban in Patients With a History of Aspirin Exacerbated Respiratory Disease
Brief Title: Trial to Determine the Safety of Oral Ifetroban in Patients With a History of Aspirin Exacerbated Respiratory Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPI-IFE-003
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Aspirin Exacerbated Respiratory Disease (AERD)
Keywords: Samster's triad; Acetylsalicylic acid triad; Widal's triad; Francis' triad; Aspirin triad; Aspirin-induced asthma and rhinitis (AIAR)
MeSH Terms: conditions — Asthma, Aspirin-Induced; Rhinitis | interventions — ifetroban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ifetroban, Oral Capsule (Active Comparator): Ifetroban, Oral Capsule; 200 mg per dose (four - 50 mg capsules), once per day on Study Days 1, 2, and 3.
  Interventions: Drug: Ifetroban, Oral Capsule
- Placebo, Oral Capsule (Placebo Comparator): Placebo, Oral Capsule; matching capsules for oral ifetroban dosing, four capsules once per day on Study Days 1, 2, and 3.
  Interventions: Drug: Placebo, Oral Capsule

INTERVENTIONS:
Drug: Ifetroban, Oral Capsule
  Arms: Ifetroban, Oral Capsule
Drug: Placebo, Oral Capsule
  Arms: Placebo, Oral Capsule

SUMMARY:
The primary objective of the study is to determine the safety of oral ifetroban compared to placebo as measured by a > 20% decrease in FEV1 compared to baseline following a dose of Investigational Medicinal Product (IMP) (Study Day 1 or 2) prior to initiation of the aspirin challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with a history of physician-diagnosed stable asthma (FEV1 of at least 1.25 liters and 60% or better than predicted* on two previous visits with no more than a 10% variation in those values, no increase in baseline dose of oral glucocorticoids for asthma for at least three months, and no history of hospitalization or emergency room visits for asthma for at least the prior six months).
2. Have a history of nasal polyposis.
3. Have a history of at least one clinical reaction to oral aspirin or other nonselective cyclooxygenase (COX) inhibitor with features of lower (cough, chest tightness, wheezing, dyspnea) and/or upper (rhinorrhea, sneezing, nasal obstruction, conjunctival itching and discharge) airway involvement.
4. Currently receiving montelukast (at least 10 mg per day, oral) or Zafirlukast (at least 20 mg twice per day, oral), with at least 1 week of therapy prior to first dose of IMP.

Exclusion Criteria:

1. Be less than 18 years of age or greater than or equal to 65 years of age.
2. Be pregnant, nursing, or planning to become pregnant.
3. Be a current tobacco smoker (defined as a daily tobacco smoker during any of the six months preceding this study or more than one instance of tobacco smoking in the last three months).
4. Use of a beta blocker in the last week.
5. Use of an antihistamine in the 48 hours prior to the first dose of IMP.
6. Use of nasal decongestants in the 48 hours prior to the first dose of IMP.
7. Use of aspirin or non-steroidal inflammatory drug (NSAID) in the last two weeks.
8. Use of zileuton in the last two weeks.
9. Have required one or more doses of ≥ 40 mg prednisone or equivalent in the last two weeks.
10. Have a history of systemic or life-threatening respiratory reaction to aspirin requiring intubation or administration of epinephrine.
11. Have a history of peptic ulcer disease, gastrointestinal bleed, or current severe gastro-esophageal reflux disease (GERD), defined as a patient currently requiring more than two total doses of medication per day to treat persistent symptoms: either more than two doses of any single medication type (antacid, proton pump inhibitor, or H2 receptor antagonist), or more than 2 types of medication per day to treat symptoms.
12. Have a history of tolerating a COX-1 blocking drug after their history of a respiratory reaction to a similar drug.
13. Have a history of cardiovascular disease including myocardial infarction, heart failure, atrial or ventricular rhythm disturbances, or angina, or a previous abnormal electrocardiogram.
14. Have a history of bleeding diathesis or use of anticoagulant or antiplatelet drugs in the last two weeks.
15. Have a history of allergy or hypersensitivity to ifetroban.
16. Have taken investigational drugs within 30 days before IMP administration.
17. Inability to understand the requirements of the study, inability to understand spoken English and abide by the study restrictions and to return for the required treatments and assessments.
18. Be otherwise unsuitable for the study, in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Scripps Clinic, San Diego, California
  - Kansas City Allergy and Asthma Associates, PA., Overland Park, Kansas
  - Allergy & Asthma Consultants of Rockland & Bergen, West Nyack, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Ifetroban, Oral Capsule: Ifetroban, Oral Capsule; 200 mg per dose (four - 50 mg capsules), once per day on Study Days 1, 2, and 3.
  Ifetroban, Oral Capsule
- Placebo, Oral Capsule: Placebo, Oral Capsule; matching capsules for oral ifetroban dosing, four capsules once per day on Study Days 1, 2, and 3.
  Placebo, Oral Capsule
Period: Overall Study
Arm/Group | Ifetroban, Oral Capsule | Placebo, Oral Capsule
Started | 14 | 5
Completed | 12 | 4
Not Completed | 2 | 1
Not completed — Inclusion or exclusion criteria not met | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ifetroban, Oral Capsule | Placebo, Oral Capsule | Total
Number analyzed (Participants) | 12 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (11.6) | 43 (13.4) | 45 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 10 | 3 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 9 | 4 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Experience a ≥ 20% Decrease in Forced Expiratory Volume in One Second (FEV1) Compared to Baseline Following a Dose of Investigational Medicinal Product (IMP) (Study Day 1 or 2) Prior to Initiation of the Aspirin Challenge
Time Frame: Study Day 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ifetroban, Oral Capsule | Placebo, Oral Capsule
Number analyzed (Participants) | 12 | 4
Participants | 0 | 0

2. Secondary Outcome: Proportion of Patients With a ≥ 25% Decrease in Peak Nasal Inspiratory Flow Rate Compared to Baseline Following a Dose of IMP (Study Day 1 or 2) Prior to Initiation of the Aspirin Challenge
Time Frame: Up to Study Day 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ifetroban, Oral Capsule | Placebo, Oral Capsule
Number analyzed (Participants) | 12 | 4
Participants | 2 | 1

3. Secondary Outcome: Proportion of Patients With a ≥ 25% Increase in Total Nasal Symptom Score (TNSS) Compared to Baseline Following a Dose of IMP (Study Day 1 or 2) Prior to Initiation of the Aspirin Challenge
Time Frame: Up to Study Day 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ifetroban, Oral Capsule | Placebo, Oral Capsule
Number analyzed (Participants) | 12 | 4
Participants | 0 | 0

4. Secondary Outcome: Incidence and Severity of Treatment-emergent Adverse Events
Time Frame: Up to Study Day 7
Population: Number of subject reporting at least one adverse event
Measure: Count of Participants; unit: Participants
Arm/Group | Ifetroban, Oral Capsule | Placebo, Oral Capsule
Number analyzed (Participants) | 12 | 4
Participants | 11 | 4

5. Secondary Outcome: Proportion of Patients Who Experience a ≥ 20% Decrease in FEV1 Compared to Baseline During the Aspirin Challenge
Time Frame: Study Day 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ifetroban, Oral Capsule | Placebo, Oral Capsule
Number analyzed (Participants) | 12 | 4
Participants | 0 | 0

6. Secondary Outcome: Proportion of Patients With a ≥ 25% Decrease in Peak Nasal Inspiratory Flow Rate (NIFR) Compared to Baseline During the Aspirin Challenge
Time Frame: Study Day 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ifetroban, Oral Capsule | Placebo, Oral Capsule
Number analyzed (Participants) | 12 | 4
Participants | 4 | 1

7. Secondary Outcome: Proportion of Patients With a ≥ 25% Increase in TNSS Compared to Baseline During the Aspirin Challenge
Time Frame: Study Day 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ifetroban, Oral Capsule | Placebo, Oral Capsule
Number analyzed (Participants) | 12 | 4
Participants | 3 | 1

8. Secondary Outcome: Amount of Rescue Medication Required During the Aspirin Challenge
Description: The amount of rescue medication required during the aspirin challenge
Time Frame: Study Day 2 and 3
Measure: Mean (Standard Deviation); unit: number of rescue medications
Arm/Group | Ifetroban, Oral Capsule | Placebo, Oral Capsule
Number analyzed (Participants) | 12 | 4
number of rescue medications | 2.9 (2.02) | 7.33 (3.79)

9. Secondary Outcome: Incidence and Severity of Asthmatic Reactions During the Treatment Period
Time Frame: Study Day 1 through 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ifetroban, Oral Capsule | Placebo, Oral Capsule
Number analyzed (Participants) | 12 | 4
Participants | 0 | 0

10. Secondary Outcome: Proportion of Patients With an Aspirin Desensitization Dose Level of 30 mg, 60 mg, 100 mg, 150 mg, and 325 mg.
Time Frame: Study Day 2 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ifetroban, Oral Capsule | Placebo, Oral Capsule
Number analyzed (Participants) | 12 | 4
Participants
  30 mg aspirin dose | 0 | 0
  60 mg aspirin dose | 5 | 2
  100mg aspirin dose | 5 | 1
  150 mg aspirin dose | 0 | 0
  325 mg aspirin dose | 0 | 0
  No Aspirin Reaction | 2 | 1

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Ifetroban, Oral Capsule | Placebo, Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4
Other Adverse Events (participants affected / at risk) | 11/12 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ifetroban, Oral Capsule (N=12) | Placebo, Oral Capsule (N=4)
Rhinnorrhea (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Forced expiratory volume decreased (Investigations) | 9 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Chest discomfort (General disorders) | 4 | 1
Eye pruritis (Eye disorders) | 3 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Conjunctivitis (Infections and infestations) | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No